CLINICAL TRIAL: NCT00085969
Title: A Phase 2, Randomized, Triple-Blind, Placebo-Controlled, Multicenter Study to Examine the Effect of Exenatide Monotherapy on Glucose Control in Subjects With Type 2 Diabetes Mellitus
Brief Title: Effect of Exenatide Monotherapy on Glucose Control in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2993-120
Record Dates: First submitted 2004-06-18; First posted 2004-06-22 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; exenatide; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- A1 - Placebo 0.04 mL twice daily (Placebo Comparator)
  Interventions: Drug: Placebo 0.04 mL twice daily
- A2 - Placebo 0.04 mL once daily (Placebo Comparator)
  Interventions: Drug: Placebo 0.04 mL once daily
- A3 - Placebo 0.08 mL once daily (Placebo Comparator)
  Interventions: Drug: Placebo 0.08 mL once daily
- B - Exenatide 10 mcg twice daily (Experimental)
  Interventions: Drug: B - Exenatide 10 mcg twice daily
- C - Exenatide 10 mcg once daily (Experimental)
  Interventions: Drug: C - Exenatide 10 mcg once daily
- D - Exenatide 20 mcg once daily (Experimental)
  Interventions: Drug: Exenatide 20 mcg once daily

INTERVENTIONS:
Drug: Placebo 0.04 mL twice daily — Subcutaneously injected, 0.04 mL, twice daily
  Arms: A1 - Placebo 0.04 mL twice daily
Drug: Placebo 0.04 mL once daily — Subcutaneously injected, 0.04 mL, once daily
  Arms: A2 - Placebo 0.04 mL once daily
Drug: Placebo 0.08 mL once daily — Subcutaneously injected, 0.08 mL, once daily
  Arms: A3 - Placebo 0.08 mL once daily
Drug: B - Exenatide 10 mcg twice daily — Subcutaneously injected, 10 mcg (0.04 mL), twice daily
  Other Names: ACC2993; synthetic exendin-4
  Arms: B - Exenatide 10 mcg twice daily
Drug: C - Exenatide 10 mcg once daily — Subcutaneously injected, 10 mcg (0.04 mL), once daily
  Other Names: ACC2993; synthetic exendin-4
  Arms: C - Exenatide 10 mcg once daily
Drug: Exenatide 20 mcg once daily — Subcutaneously injected, 20 mcg (0.08 mL), once daily
  Other Names: ACC2993; synthetic exendin-4
  Arms: D - Exenatide 20 mcg once daily

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a 28-day regimen of exenatide (AC2993), given as a monotherapy to subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Subject has type 2 diabetes mellitus treated with diet and exercise modification alone or in combination with one oral antidiabetic agent for no longer than 4 years.

Exclusion Criteria:

* Subject has a clinically significant history or presence of any of the following conditions: (a) Hepatic disease, (b) Renal disease, (c) Central nervous system disease, (d) Gastrointestinal disease (e) Pulmonary disease (f) Hematologic disease.
* Subject is currently treated with any of the following excluded medications: (a) Metformin/sulfonylurea combination therapy (b) Thiazolidinediones (c) Insulin as outpatient therapy (d) Regular use of drugs that directly affect gastrointestinal motility (e) Regular use of systemic corticosteroids by oral, intravenous (IV), or intramuscular (IM) route, or potent, inhaled, intrapulmonary, or intranasal steroids known to have a high rate of systemic absorption (f) Regular use of medications with addictive potential such as opiates, narcotics and tranquilizers (g) Antineoplastic agents (h) Transplantation medications (i) Prescription weight-loss medications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2003-09; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c (glycosylated hemoglobin) from Baseline to Day 28 | Baseline, Day 28
  Change in HbA1c from Baseline Visit 3 (Day 1) to study termination (Day 28)

SECONDARY OUTCOMES:
Change in serum fructosamine concentration from Baseline to Day 14 and to Day 28 | Baseline, Day 14, Day 28
  Change in serum fructosamine concentration from Baseline Visit 3 (Day 1) to Visit 4 (Day 14) and to study termination (Day 28)
Change in body weight from Baseline to Day 14 and to Day 28 | Baseline, Day 14, Day28
  Change in body weight from Baseline Visit 3 (Day 1) to Visit 4 (Day 14) and to study termination (Day 28)
Change in fasting plasma glucose concentration from Baseline to Day 14 and to Day 28 | Baseline, Day 14, Day 28
  Change in fasting plasma glucose concentration from Baseline Visit 3 (Day 1) to Visit 4 (Day 14) and to study termination (Day 28)
Change in postprandial blood glucose concentrations from Baseline to Day 28 | Baseline, Week 28
  Change in postprandial blood glucose concentrations from Baseline Visit 3 (Day 1) to study termination (Day 28)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - The Whittier Institute for Diabetes, La Jolla, California
  - VA Medical Center, San Diego, California
  - MedStar Research Institute, Washington D.C., District of Columbia
  - Internal Medicine Associates, Department of Research, Fort Myers, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Innovative Research of West Florida, Largo, Florida
  - Henry Ford Health System, Detroit, Michigan
  - Grand Rapids Associated Internists, Grand Rapids, Michigan
  - Radiant Research, Inc., St Louis, Missouri
  - Internal Medicine Associates, Bozeman, Montana
  - Mercury Street Medical Group, Butte, Montana
  - Lovelace Scientific Resources, Las Vegas, Nevada
  - Rochester Clinical Research, Inc., Rochester, New York
  - Metrolina Medical Research, Charlotte, North Carolina
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - Radiant Research, Columbus, Ohio
  - Smith Clinic Research, Marion, Ohio
  - Radiant Research, Portland, Oregon
  - Philadelphia Health Associates - Adult Medicine, Philadelphia, Pennsylvania
  - Diabetes and Glandular Disease Research Associates, San Antonio, Texas
  - S.A.M. Clinical Research Center, San Antonio, Texas
  - McGuire VA Medical Center, Richmond, Virginia
  - Rockwood Clinic, Spokane, Washington

REFERENCES:
- [Derived] Nelson P, Poon T, Guan X, Schnabel C, Wintle M, Fineman M. The incretin mimetic exenatide as a monotherapy in patients with type 2 diabetes. Diabetes Technol Ther. 2007 Aug;9(4):317-26. doi: 10.1089/dia.2006.0024. PMID 17705687